CLINICAL TRIAL: NCT01399008
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of MBX-102 in Combination With Allopurinol in Gout Patients With an Inadequate Hypouricemic Response to Allopurinol Alone
Brief Title: Safety/Efficacy Study to Evaluate of MBX-102 in Combination With Allopurinol in Gout Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M102-21123
Record Dates: First submitted 2011-07-13; First posted 2011-07-21 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Gout
Keywords: Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — arhalofenate; Allopurinol; Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arhalofenate 400 mg (Experimental): Arhalofenate 400 mg plus allopurinol 300 mg
  Interventions: Drug: Arhalofenate; Drug: Allopurinol; Drug: Colchicine
- Arhalofenate 600 mg (Experimental): Arhalofenate 600 mg plus allopurinol 300 mg
  Interventions: Drug: Arhalofenate; Drug: Allopurinol; Drug: Colchicine
- Allopurinol (Active Comparator): Placebo plus Allopurinol 300 mg
  Interventions: Drug: Allopurinol; Drug: Colchicine; Drug: Placebo

INTERVENTIONS:
Drug: Arhalofenate — Arhalofenate 400 and 600 mgs over-encapsulated tablets once daily for 4 weeks or Allopurinol 300 mg once daily for 4 weeks
  Arms: Arhalofenate 400 mg; Arhalofenate 600 mg
Drug: Allopurinol — Allopurinol 300 mg as active comparator
Drug: Colchicine — 0.6 mg colchicine daily as flare prophylaxis
Drug: Placebo — Placebo
  Arms: Allopurinol

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of MBX-102 in combination with allopurinol compared to allopurinol alone when administered orally once a day for four weeks to gout patients with an inadequate hypouricemic response to allopurinol alone.

ELIGIBILITY:
Inclusion Criteria:

1. Known gout patients (per criteria of the American Rheumatism Association for the classification of the acute arthritis of primary gout

   1. Patients who have been taking at least 200 mg/day of allopurinol as the sole ULT for at least two weeks with a sUA of ≥ 6.5 mg/dL and ≤ 12 mg/dL at screening and ≥ 6.0 mg/dL and ≤ 12 mg/dL at Week -1 (Visit 2) randomization visit.

      -OR -
   2. Patients who are not on ULT or are taking allopurinol < 200 mg/day must have a sUA ≥ 8.0 mg/dL and ≤ 12 mg/dL at screening and ≥ 6.0 mg/dL and ≤ 12 mg/dL at Week -1 (Visit 2) randomization visit.
2. Male or female, 18-75 years of age at screening
3. All female patients must be surgically sterile or post-menopausal (at least 45 years of age with no history of menses for at least 2 years; or any age with no history of menses for at least six months and serum FSH ≥ 40 mIU/mL) or have a partner who has undergone vasectomy or must agree to use two medically accepted methods of contraception including a barrier method (see the list in Appendix 4) for the entire duration of the study unless she reports complete sexual abstinence.
4. Female patients must not be pregnant or lactating.
5. Male patients with a female partner of child-bearing potential must agree to use condoms or the partner must use a medically acceptable method of contraception for the entire duration of the study.
6. Estimated creatinine clearance (CrCl) by Cockcroft-Gault method ≥ 60 mL/min at screening
7. Serum creatinine value ≤ 1.1 mg/dL in females and ≤ 1.3 mg/dL in males
8. Liver function tests ≤ 1.5X ULN for AST, ALT and T-bilirubin, ≤ 2X ULN for ALP, ≤ 3X ULN for GGT; and ≤ 3X ULN for CK
9. All other clinical laboratory parameters must be within normal limits or considered not clinically significant for participation in this study.
10. Electrocardiogram (ECG) must be normal, or if abnormal, considered not clinically significant for participation in this study.
11. Systolic blood pressure ≤ 160 mm Hg and diastolic blood pressure ≤ 90 mm Hg; known hypertensive patients controlled with medications other than thiazide diuretics (blood pressure [BP] reading as above) may be included

Exclusion Criteria:

1. Treatment with any ULT other than allopurinol (e.g., probenecid, benzbromarone, febuxostat, or pegloticase) within 30 days of the Screening Visit
2. Known or suspected secondary hyperuricemia (e.g. due to myeloproliferative disorder, or organ transplant)
3. Diagnosis of xanthinuria
4. History of documented or suspected kidney stones
5. Known infection with HIV or history of viral hepatitis type B or C
6. History of illicit drug or alcohol abuse within 1 year of screening
7. History of significant pulmonary disease, upper GI bleeding, documented peptic ulcer disease (unless known H. pylori infection treated successfully without recurrence), or nephrotic syndrome within three years of screening
8. History of stroke, TIA, acute MI, congestive heart failure (NYHA Class II-IV), angina pectoris, coronary intervention procedure (including but not limited to angioplasty, stent placement, coronary revascularization), lower extremity bypass procedure, systemic or intracoronary fibrinolytic therapy within five years of screening
9. Malignancy (except treated basal cell carcinoma) within five years of screening
10. BMI > 42 kg/m2
11. Current or expected requirement for anticoagulant therapy (except for aspirin ≤ 325 mg/day)
12. Rheumatoid arthritis or other autoimmune disease requiring ongoing treatment
13. Current or expected treatment with potent CYP3A4 inhibitors (See Appendix 6), cytotoxic agents (azathioprine, mercaptopurine, cyclosporine, cyclophosphamide, etc.), ranolazine, digoxin, theophylline, sulphonylureas, thiazolidinediones, diuretics, atypical antipsychotic agents, ampicillin, amoxicillin or phenytoin
14. Chronic treatment with NSAIDs (use to treat acute flares are permitted).
15. Current or expected treatment with systemic corticosteroids (except topical, ophthalmic, intra-articular, or inhaled at a dose < 1600 μg/day) other than to treat acute flare
16. Known hypersensitivity to allopurinol, colchicine, or aspirin
17. Treatment with any other investigational therapy within the 30 days prior to screening, or patients who received at least one dose of study drug while enrolled in any previous or concomitant MBX-102 trial
18. Any other condition that compromises the ability of the patient to provide informed consent or to comply with the objectives and procedures of this protocol, as judged by the investigator and/or medical monitor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (16):
  - Lincoln, California
  - Los Angeles, California
  - Palo Alto, California
  - Boca Raton, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Honolulu, Hawaii
  - Baltimore, Maryland
  - Brockton, Massachusetts
  - St Louis, Missouri
  - Hartsdale, New York
  - New York, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - San Antonio, Texas
  - West Jordan, Utah
- Canada (7):
  - Burnaby, British Columbia
  - St. John's, Newfoundland and Labrador
  - London, Ontario
  - Sarnia, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
  - Mirabel, Quebec
- Tbilisi, Georgia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Upon completion of screening all patients will enter into a 3-week run-in/stabilization period starting at Week -3 (Visit 1). During this phase, all patients will take allopurinol 300 mg once daily. In addition, patients will be given colchicine 0.6 mg once daily until the final study visit as prophylaxis to prevent potential gout flares.
Groups:
- Placebo: Placebo plus Allopurinol 300 mg
Period: Overall Study
Arm/Group | Arhalofenate 400 mg | Arhalofenate 600 mg | Placebo
Started | 35 | 32 | 33
Completed | 32 | 27 | 31
Not Completed | 3 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arhalofenate 400 mg | Arhalofenate 600 mg | Placebo | Total
Number analyzed (Participants) | 35 | 32 | 33 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (10.9) | 50.6 (10.2) | 50.4 (11.0) | 51.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1
  Male | 35 | 32 | 32 | 99

OUTCOME MEASURES:

1. Primary Outcome: Serum Uric Acid
Description: Percent change from baseline in serum uric acid in Per Protocol population
Time Frame: Percent change from baseline in serum uric acid at Week 4
Population: Per Protocol population (all randomized patients who received at least 1 dose of blinded study drug, had at least 1 post-treatment evaluation, had not violated any major entry criterion likely to confound an efficacy analysis and had not deviated significantly from the protocol between enrollment and study completion).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Arhalofenate 400 mg | Arhalofenate 600 mg | Placebo
Number analyzed (Participants) | 34 | 30 | 31
percent change | -16.0 (20.9) | -9.9 (17.1) | -9.5 (19.0)

ADVERSE EVENTS:
Time Frame: 6 weeks (Treatment/Post Treatment Periods)
Groups:
- Arhalofenate 400 mg Plus Allopurinol 300 mg: Arhalofenate 400 mg plus allopurinol 300 mg (Safety Population)
- Arhalofenate 600 mg Plus Allopurinol 300 mg: Arhalofenate 600 mg plus allopurinol 300 mg (Safety Population)
- Placebo Plus Allopurinol 300 mg: Placebo plus allopurinol 300 mg (Safety Population)
Arm/Group | Arhalofenate 400 mg Plus Allopurinol 300 mg | Arhalofenate 600 mg Plus Allopurinol 300 mg | Placebo Plus Allopurinol 300 mg
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 10/35 | 6/32 | 9/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arhalofenate 400 mg Plus Allopurinol 300 mg (N=35) | Arhalofenate 600 mg Plus Allopurinol 300 mg (N=32) | Placebo Plus Allopurinol 300 mg (N=33)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Gout flare (Renal and urinary disorders) | 10 | 2 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication requires the prior written consent of the Sponsor. The Principal Investigator must provide the Sponsor the opportunity to review any proposed abstracts, manuscripts or presentations that relate to any research or clinical results at least 30 days prior to its intended submission for publication.